CLINICAL TRIAL: NCT00820443
Title: Ceramic on Metal Total Hip Replacement System IDE: A Non-Randomized, Multi-center, Historically Controlled Safety and Efficacy Study (Protocol Number:06-LJH-002)
Brief Title: Ceramic on Metal Total Hip Replacement System Multi-Center,Investigational Device Exemption Clinical Trial
Acronym: COM
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: not move forward with the commercialization of this product based on marketing needs and there is not a known safety issue or concern
Sponsor: MicroPort Orthopedics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06LJH002
Record Dates: First submitted 2009-01-08; First posted 2009-01-12 (Estimated); Results first posted 2015-09-30 (Estimated); Last update posted 2015-09-30 (Estimated); Status verified 2015-08

CONDITIONS: Total Hip Replacement System

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ceramic on metal prosthesis (Experimental): Ceramic on metal prosthesis
  Interventions: Device: Ceramic on metal prosthesis

INTERVENTIONS:
Device: Ceramic on metal prosthesis — Ceramic femoral head with a metal acetabular component

SUMMARY:
The purpose of this study is to demonstrate non-inferiority of the Ceramic on Metal Total Hip when compared to a TRANSCEND® historical control group of patients with primary total hip replacement.

DETAILED DESCRIPTION:
This investigational device study is a non-randomized, non-inferiority, multi-center, historically controlled study. The primary objective will be evaluated at the primary endpoint (24 months) by the primary efficacy and safety measures that define patient success. The proportion of patient success will determine whether the primary objective has been met (study success).

The investigational device will be compared to a historical control comprised of patients from the TRANSCEND® Ceramic on Ceramic IDE study. This comparison will be made using all primary and secondary measures. However, only primary measures will be used to determine study success.

ELIGIBILITY:
Inclusion Criteria:

1. Must be 18 years of age or older at the time of enrollment,
2. Patient is skeletally mature,
3. Evidence of a signed and dated informed consent document indicating that the patient has been informed of all pertinent aspects of the study,
4. Patient agrees to comply with this protocol, including participating in required follow-up visits at the investigational site and completing study questionnaires, (i.e. patient's reasonable driving distance to assure study follow-up and completion)
5. Investigator determines patient is a suitable candidate for primary total hip replacement,
6. Body Mass Index (BMI) of <40,
7. Preoperative Harris Hip Score (HHS) < 70 points as calculated on the Pre-screening Qualification Form and verified by the Sponsor,
8. Have a diagnosis of degenerative joint disease of the hip.

Exclusion Criteria:

1. Previous total hip replacement, hemi-arthroplasty, or fusion on the ipsilateral side,
2. Patients with a previous Girdlestone procedure,
3. Patient has a known metal allergy to any component of the investigational device (e.g.cobalt, chromium, titanium or ceramics),
4. Patient has had a total knee arthroplasty of either leg,
5. Patient has vascular insufficiency, muscular atrophy, or neuromuscular disease in the affected limb (based on the Investigator's discretion),
6. Patients with congenital disorder or deformity not adequately addressed by hip replacement or has sufficient anatomic variance or remodeling of the hip joint that may place the patient at risk for mechanical failure or that requires a structural bone graft (based on the Investigator's discretion),
7. Patients with severe instability or deformity of the ligaments or surrounding soft tissues that would preclude stability of the implant (based on the Investigator's discretion),
8. Patients with Charcot or neuropathic arthropathy, or neuromuscular disease or any other condition that would interfere with patient self-assessment or pain, the function or quality of life required for patient reported outcomes during the study (based on the Investigator's discretion),
9. Patient, male or postmenopausal female, with a history of metabolic bone disease, as defined by the following:

   * Osteoporosis where the patient is currently taking prescription medications that increase bone-mineral density (e.g. Fosamax, Didronel), or
   * Patient was previously diagnosed with a metabolic bone disease (e.g. Paget's disease or osteomalacia), or
   * Patient has any other metabolic bone disease to a degree that the investigator determines that a THR would be contraindicated,
10. Active malignancy,
11. Patient has an active infection (e.g. hepatitis, AIDS, ARC or is HIV positive)- systemic or at the site of intended surgery,
12. Clinical diagnosis of renal insufficiency where renal function is abnormal and incapable of sustaining essential bodily functions. (e.g. as reported by KRONOS lab BUN, Creatinine and estimated glomerular filtration rate (GFR <15 mL/min/1.73 m2)
13. Currently participating in any investigational studies not related to this study's preoperative or postoperative care,
14. Patient has a mental illness or belongs to a vulnerable population (e.g., is a prisoner or a severe drug abuser, or is developmentally disabled) such that his or her ability to provide informed consent or comply with follow-up requirements is compromised,
15. Patient is pregnant or interested in becoming pregnant in the next 2 years, (Due to the required x-rays for the study),
16. Other severe acute or chronic medical condition that may interfere with the interpretation of the study results, in the judgment of the investigator, which would make the patient inappropriate for entry into this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 253 (Actual)
Dates: Start 2007-06; Primary Completion 2013-06 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- St. Vincent's Hospital, Los Angeles, California, United States

REFERENCES:
- [Result] National Kidney Foundation. K/DOQI clinical practice guidelines for chronic kidney disease: evaluation, classification, and stratification. Am J Kidney Dis. 2002 Feb;39(2 Suppl 1):S1-266. No abstract available. PMID 11904577

RESULTS

PARTICIPANT FLOW:
Groups:
- Ceramic on Metal Prosthesis: Ceramic on metal prosthesis
  Ceramic on metal prosthesis: Ceramic femoral head with a metal acetabular component Ceramic large head with monoblock or modular acetabular component
Period: Pre-Op
Arm/Group | Ceramic on Metal Prosthesis
Started | 253
Completed | 253
Not Completed | 0
Period: Op
Arm/Group | Ceramic on Metal Prosthesis
Started | 253
Completed | 253
Not Completed | 0
Period: Immediately
Arm/Group | Ceramic on Metal Prosthesis
Started | 253
Completed | 248
Not Completed | 5
Period: 3 Month
Arm/Group | Ceramic on Metal Prosthesis
Started | 253
Completed | 244
Not Completed | 9
Period: 6 Month
Arm/Group | Ceramic on Metal Prosthesis
Started | 253
Completed | 233
Not Completed | 20
Period: 12 Month
Arm/Group | Ceramic on Metal Prosthesis
Started | 250
Completed | 226
Not Completed | 24
Period: 24 Month
Arm/Group | Ceramic on Metal Prosthesis
Started | 245
Completed | 202
Not Completed | 43

BASELINE CHARACTERISTICS:
Arm/Group | Ceramic on Metal Prosthesis
Number analyzed (Participants) | 253
Age, Continuous [Mean (Standard Deviation); unit: years]
  Female | 60.8 (12.9)
  Male | 60.3 (13.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 128
  Male | 125
BMI [Mean (Standard Deviation); unit: kg/m^(2)]
  Female | 28.2 (5.2)
  Male | 29.1 (4.6)
Height [Mean (Standard Deviation); unit: Inches]
  Female | 64.2 (2.4)
  Male | 70.4 (3.0)
Weight [Mean (Standard Deviation); unit: lbs]
  Female | 164.7 (31.1)
  Male | 205.4 (37.3)
Diagnosis [Number; unit: participants]
  Osteo/degenerative arthritis | 216
  Post-traumatic Arthritis | 4
  Avascular necrosis | 25
  Rheumatoid Arthritis | 3
  Congenital Hip Dysplasia | 5

OUTCOME MEASURES:

1. Primary Outcome: Primary Endpoint/Measures: Success at 24 Months
Description: The patient success definition is measured at the 24 month interval by the following:
  * Harris Hip Score (HHS) of > 80 • < 2mm radiolucency (width) in any Gruen (stem) or DeLee/Charnley (cup) zone and no more than mild pain.
  * No revision or removal of any part of the device for aseptic reasons prior to or on day 730 following the index surgical procedure.
  A patient must meet all three criteria in the definition to be considered a success. A patient who does not meet all three criteria will be deemed a failure.
  The Harris hip score, is used to measure the outcome of total hip arthroplasty. Eight sections on the HIP are rated by the patient: pain, distance walked, activities, public transportation, support, limp, stairs and sitting. Total scores are out of 100 and grouped as follows: 90 - 100 Excellent,80 - 90 Good,70 - 79 Fair,60 - 69 Poor.< 60 Failed.Any score above 60 is acceptable, although the higher the score, the better the patient's overall adjustment after the surgery
Time Frame: 24 Month
Population: Patients with Harris Hip Score (HHS) of > 80 Because there isn't complete radiographic data,the composite primary outcome is not analyzed at 24 month as in protocol. Only the number of patients who has HHS score greater that 80 is entered.Due to missing values/assessments/data, not all of the participants were evaluated at 24 months, only 197.
Measure: Number; unit: participants
Arm/Group | Ceramic on Metal Prosthesis
Number analyzed (Participants) | 197
participants | 163

2. Secondary Outcome: The Secondary Measures of the UCLA Functional Assessments
Description: UCLA: University of California LosAngeles Activity Score
  UCLA score is a validated scoring system for hip replacement outcome, The single item UCLA scale asks patients to rate their activity level from 1 to 10, with 1 defined as "no physical activity" and 10 defined as "regular participation in impact sports". The score is the higher the better.
Time Frame: 24 months
Population: Due to missing values/assessments/data, not all of the participants were evaluated at 24 months, only 177 participants were evaluated at 24 months.
Measure: Mean (Standard Deviation); unit: units on a scale (10 points)
Arm/Group | Ceramic on Metal Prosthesis
Number analyzed (Participants) | 177
units on a scale (10 points) | 6.8 (1.7)

3. Secondary Outcome: WOMAC Raw Total Score
Description: The Western Ontario and McMaster Universities Arthritis Index (WOMAC) is a widely used, proprietary set of standardized questionnaires used by health professionals to evaluate the condition of patients with osteoarthritis of the knee and hip, including pain, stiffness, and physical functioning of the joints The WOMAC measures five items for pain (score range 0-20), two for stiffness (score range 0-8), and 17 for functional limitation (score range 0-68). Physical functioning questions cover everyday activities such as stair use, standing up from a sitting or lying position, standing, bending, walking, getting in and out of a car, shopping, putting on or taking off socks, lying in bed, getting in or out of a bath, sitting, and heavy and light household duties Higher scores on the WOMAC indicate worse pain, stiffness, and functional limitations (range is 0-96).
Time Frame: 24 months
Population: Due to missing values/assessments/data, not all of the participants were evaluated at 24 months, only 175 participants were evaluated at 24 months.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ceramic on Metal Prosthesis
Number analyzed (Participants) | 175
units on a scale | 5.3 (11.1)

4. Secondary Outcome: Metal Ion Analysis (Unilateral Only):Serum Cobalt
Description: Serum cobalt and chromium are recommended as the optimal tests for evaluation of joint implant wear, patients with CoM implants have elevated serum chromium and cobalt concentrations. Clinically important implant wear is indicated when serum chromium exceeds 15 ng/mL and cobalt exceeds 10 ng/mL; these symptomatic patients are likely to have significant implant deterioration. serum cobalt and chromium are highest in the first year after implant. In subsequent years, and after run-in wear (initial wear of a hip implant that produces the greatest amount of metal ion release), cobalt and chromium concentrations decline, then reach steady state around 3 years after implant.
Time Frame: 24 months
Population: Only Unilateral participants were collected the Metal Ion data, and due to missing values/assessments/data, not all of the unilateral participants had Metal Ion data at 24 months, only 44 of them were evaluated.
Measure: Mean (Standard Deviation); unit: ug/L
Arm/Group | Ceramic on Metal Prosthesis
Number analyzed (Participants) | 44
ug/L | 1.06 (0.12)

5. Secondary Outcome: Metal Ion Analysis; Unilateral Only; Serum Chromium
Description: as for outcome 4
Time Frame: 24 months
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: ug/L
Arm/Group | Ceramic on Metal Prosthesis
Number analyzed (Participants) | 44
ug/L | 0.79 (0.12)

ADVERSE EVENTS:
Time Frame: The period includes all the time with a date of surgery on or before the date of database closure.
Description: The AE for all enrolled procedures with a date of surgery on or before the date of database closure are included. n/N, n=number of procedure with a specific complication, N is the total number of procedure implanted and evaluated (N=253). Both AE and SAE are separated and re-coded (MedDRA18.0). For other AE, only >=5% frequency are reported.
Arm/Group | Ceramic on Metal Prosthesis
Serious Adverse Events (participants affected / at risk) | 22/253
Other Adverse Events (participants affected / at risk) | 85/253
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ceramic on Metal Prosthesis (N=253)
Anemia (Blood and lymphatic system disorders) | 1
Atrial Fibrillation (Cardiac disorders) | 1
Osteonecrosis (Vascular disorders) | 1
Carcinoid tumor of the stomach (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cellulitis (Infections and infestations) | 1
Abscess Neck (Infections and infestations) | 1
Intermittent Claudication (Vascular disorders) | 1
Intervertebral disc operation (Surgical and medical procedures) | 1
Myocardial infarction (Vascular disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Ovarian Cancer (Reproductive system and breast disorders) | 1
Pancreatic carcinoma (Gastrointestinal disorders) | 1
Pneumonia (Infections and infestations) | 1
Retroperitoneal Haemorrhage (Gastrointestinal disorders) | 1
Hip arthroplasty (Surgical and medical procedures) | 1
Seizure (Nervous system disorders) | 1
Cardiac arrest (Cardiac disorders) | 1
Subcutaneous abscess (Skin and subcutaneous tissue disorders) | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 1
Wound infection (Infections and infestations) | 1
Surgical failure (General disorders) | 1
Chest Pain (General disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ceramic on Metal Prosthesis (N=253)
Anemia (Blood and lymphatic system disorders) | 27
Pain in Hip (Musculoskeletal and connective tissue disorders) | 22
Trochanteric bursitis (Musculoskeletal and connective tissue disorders) | 21
Knee Pain (Musculoskeletal and connective tissue disorders) | 15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days